CLINICAL TRIAL: NCT04611503
Title: PIGMENT - PDE6A Gene Therapy for Retinitis Pigmentosa
Brief Title: PDE6A Gene Therapy for Retinitis Pigmentosa
Acronym: Pigment
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: STZ eyetrial (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RDC-PDE6A-01
Record Dates: First submitted 2020-05-20; First posted 2020-11-02 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subretinal injection of rAAV.hPDE6A (Experimental): Single subretinal injection of rAAV.hPDE6A
  Interventions: Drug: subretinal injection of rAAV.hPDE6A

INTERVENTIONS:
Drug: subretinal injection of rAAV.hPDE6A — The first 3 patients (C1) will receive the intermediate dose 1x1010 vg. After injection of the 3rd patient of C1, the DMC will give a go/no go decision. If 'nogo', a lower dose (5x109 vg) will be given to the next group of 3 patients (C2). The DMC will give a go/no go decision. In case of a "go" decision, 3 further patients (C3) will be treated with the same dose. In the case of a no-go decision, the next dose will be the minimal dose 1x109 vg. In case of a 'go' decision of the DMC after the third patient, the next 3 patients will receive a subretinal injection of vector at the highest dose 5x1010 vg. The DMC will give a go/no go decision after review of all safety data available at D30 of cohort 2. If safety data is considered favourably by the DMC, then 3further patients (cohort 3) will be treated with the same dose (5x1010 vg). Should any safety concerns arise, the last three patients (cohort 3) will receive the intermediate dose (1x1010 vg).
  Other Names: Gene therapy

SUMMARY:
The PDE6A gene encodes a subunit of the rod phosphodiesterase. The loss of this enzyme function leads to a chronically elevated cGMP level which causes an increased calcium inflow into the cell and thereby the hyperactivation of cell death pathways. The goal of the PIGMENT study is to develop, produce and investigate a recombinant adeno-associated viral (AAV) gene transfer vector for the curative therapy of PDE6A-linked retinitis pigmentosa in patients, in order to counteract their disease progression and to stop further impairment of visual function. The vector is given with a single subretinal injection.

DETAILED DESCRIPTION:
"PIGMENT - Subretinal PDE6A gene therapy for retinitis pigmentosa" is an open mono-center, phase I/IIa trial with fellow-eye comparison.

The study begins with a detailed preliminary examination (Screening), comprises a total of 13 visits and ends after one year. In between, after the gene therapy injection (injection of the vector under the retina with one of four doses), regular controls are carried out at the Center for Ophthalmology Tübingen. Monitoring will be contimued after the first year, once a year two, three, four and five years after the injection. The study will take place exclusively at the Center for Ophthalmology in Tübingen and involves nine patients.

All patients participating in this study receive treatment, i.e. there is no placebo or sham treatment group. A 30-day safety distance is maintained between each patient and each group. An independent committee will decide, after each injection of three patients, which dose the following three patients will receive.

Patients can benefit from the treatment by slowing or stopping the loss of the rods and allowing them to function to a certain extent. Therefore, a possible benefit for patients may be that the vision problems will be improved by gene therapy. Such improvements could improve the overall quality of life and well-being. However, as no experience with gene therapy for retinitis pigmentosa in humans has yet been gained, we cannot promise any improvement. Within the scope of this study, patients will be given particularly intensive care and psychological support will also be offered in order to do everything for the patient's well-being and health during the study.

Time Schedule: Start of trial Q3/2019 (FPFV), end of recruitment Q3/2020, end of trial Q4/2025 (LPLV), duration of trial per patient: one year with four years of follow-up. The final study report will be prepared after completion of the four year follow-up period (5 years after treatment).

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of retinitis pigmentosa
* confirmed mutation in PDE6A gene
* ≥ 18 years of age
* visual acuity ≥ 20/400
* no infection with Human Immundeficiency Virus (HIV)
* negative pregnancy test in women with childbearing potential (a woman who is two years post-menopausal or surgically sterile is not considered to be of childbearing potential)
* Male patients must agree to use condoms during the first 6 months post treatment.
* Female patients of childbearing potential must agree to use an effective method of birth control during the first 6 months post treatment.
* ability to understand and willingness to consent to study protocol

Exclusion Criteria:

Ocular (study eye & fellow eye)

* additional interfering ocular conditions with impact on study results (e.g. ocular opacity and advanced cataract, uveitis, amblyopia)
* recent (6 months) ocular surgery, intravitreal or subretinal implantation of a medical device
* disease causing mutations in another known retinitis pigmentosa gene
* ocular infection with herpes simplex virus in medical history
* history of ocular malignancies
* disorders of the internal retina (e.g. retinal detachment in the patients history)
* glaucoma defined as damage of the optic nerve
* vascular retinal occlusion
* diabetic patients suffering from retinopathy and/or macula edema
* any other retinopathy due to other diseases e.g. (but not limited to) arterial hypertension, trauma or acquired inflammatory diseases (uveitis serology), contraindication to pharmacological mydriasis (e.g. history of angle block glaucoma)
* absence of visual function on the contralateral eye Systemic
* systemic conditions (e.g. coronary heart disease, autoimmune disorders) which may affect study participation or outcome measures
* History of poorly controlled Diabetes Mellitus type 1 or type 2
* systemic illness or medically relevant abnormal laboratory values in blood analysis including renal and hepatic functions at inclusion
* patients treated with oral corticoids within 14 days prior inclusion
* current or recent participation in other study/or administration of biologic agent within the last three months
* known sensitivity to any compound used in the study
* contraindications to systemic immunosuppression
* contraindications in view of the planned surgery (e.g. but not limited to anaemia Hb<10g/dl, coagulopathy with PT/PTT >1,5 fold upper limit, hypertension with values above 180 mmHg systolic and 110 mmHg diastolic) including intolerance and contraindications to general anaesthesia
* intolerance to contrast agents used for diagnostic methods like angiography with fluoresceine or indocyanine green (e.g. but not limited to hyperthyroidism, hepatic insufficiency)
* subject/partner of childbearing potential unwilling to use adequate contraception for four months
* nursing or pregnant women
* any other cause that, in the investigator's opinion, renders potential subjects not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Slit lamp examination | 1 year + 4 years follow-up
  to determine possibly occurring ocular inflammation and to observe if there are any treatment effects
Fundus biomicroscopy to determine possibly occurring ocular inflammation and to observe if there are any treatment effects | 1 year + 4 years follow-up
  To determine possibly occurring ocular inflammation and to observe if there are any treatment effects
Angiography | 1 year + 4 years follow-up
  To determine possibly occurring ocular inflammation and to observe if there are any treatment effects

SECONDARY OUTCOMES:
Visual acuity | 1 year + 4 years follow-up
  To determine any therapy effects concerning visual acuity
Contrast sensitivity | 1 year + 4 years follow-up
  To determine any therapy effects concerning the contrast sensitivity
Visual field | 1 year + 4 years follow-up
  To determine any therapy effects concerning the visual field
Colour vision | 1 year + 4 years follow-up
  To determine any therapy effects concerning colour vision
Pupillography | 1 year + 4 years follow-up
  To determine any therapy effects concerning pupil reaction
Electrophysiology | 1 year + 4 years follow-up
  To determine any therapy effects concerning the electrophysiology

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Fischer, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- Universitätsklinikum Tübingen, Department für Augenheilkunde, Tübingen, Germany

REFERENCES:
- [Derived] Seitz IP, Wozar F, Ochakovski GA, Reichel FF, Korte S, Korbmacher B, Wilhelm B, Susskind D, Bartz-Schmidt KU, Fischer MD, Peters T; RD Cure Consortium. Ocular Safety and Toxicology of Subretinal Gene Therapy With rAAV.hPDE6A in Nonhuman Primates. Transl Vis Sci Technol. 2025 Jan 2;14(1):29. doi: 10.1167/tvst.14.1.29. PMID 39878701